CLINICAL TRIAL: NCT06800027
Title: SALSA (Health, Food and Sociability): Community Networks for Healthy Eating, Autonomy, and Social Interaction
Acronym: SALSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Fundació Alícia (Unknown)
Responsible Party: Principal Investigator, Anna Ruiz Comellas, PHD, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23/285-P
Record Dates: First submitted 2025-01-24; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Depression; Anxiety; Social Support (formal and Informal); Quality of Life (QOL); Loneliness; Malnutrition
Keywords: Loneliness; Depression; Anxiety; Social support; Quality of life
MeSH Terms: conditions — Depression; Anxiety Disorders; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will dine at a selected and trained restaurant twice a week for 4 months (from March to June 2024). A facilitator will accompany the participants to the restaurant and supervise them. Once a month, a healthy habits and meal supplementation workshop will be held at the senior citizens' centre. Participants will not be required to pay for the meals at the restaurant or for participation in the workshops.
  In order for the restaurant to provide appropriate services tailored to the users' needs, training will be conducted by professionals from the Alicia Foundation on how to manage the nutrition of elderly individuals and other participants in the study according to their dietary needs.
  Interventions: Other: SALSA group intervention: Going to lunch at the restaurant in a group and attending healthy eating workshops.
- Control grup (No Intervention): The control group will receive standard care at their Primary Care Centre.

INTERVENTIONS:
Other: SALSA group intervention: Going to lunch at the restaurant in a group and attending healthy eating workshops. — The intervention group will dine at a selected and trained restaurant twice a week for 4 months (from March to June 2024). A facilitator will accompany the participants to the restaurant and supervise them. Once a month, a healthy habits and meal supplementation workshop will be held at the senior citizens' centre. Participants will not be required to pay for the meals at the restaurant or for participation in the workshops. The control group will receive standard care at their Primary Care Centre.
  In order for the restaurant to provide appropriate services tailored to the users' needs, training will be conducted by professionals from the Alicia Foundation on how to manage the nutrition of elderly individuals and other participants in the study according to their dietary needs.
  Arms: Intervention group

SUMMARY:
Antecedents: Unwanted loneliness is associated with an increased risk of anxiety, depression, social isolation, and malnutrition. The SALSA project aims to establish mechanisms and create an ecosystem that enables healthcare and social services to prescribe meals at pre-trained local restaurants. The goal is to encourage socialisation and simultaneously ensure a diet tailored to the user's needs, without stigmatisation, new infrastructure, or additional staffing.

Hypotheses: Individuals experiencing unwanted loneliness with a risk of anxiety, depression, and malnutrition will improve their emotional and nutritional status, social support, and quality of life if they dine at a restaurant in a group, accompanied by a facilitator, twice a week.

Objectives: To assess whether dining at a restaurant twice a week in a group, accompanied by a facilitator, and participating in healthy eating workshops improves the emotional and nutritional status, social support, and quality of life of individuals experiencing unwanted loneliness.

Methodology:

Design: Randomised clinical trial with two groups. Inclusion Criteria: Autonomous individuals experiencing challenges related to living alone (Z60), at risk of malnutrition or emotional disorders, with a score of ≥14 and <28 on the Beck Depression Inventory (BDI-II), ≥10 on the Generalised Anxiety Disorder scale (GAD-7), or ≥32 on the DUKE-UNC-11 Social Support Scale. Participants must be able to attend follow-ups over eight months, read and write in Spanish or Catalan, and dine at a restaurant twice a week.

Measurements: Sociodemographic variables, assessments of depression, anxiety, social support, quality of life, and clinical variables such as weight, height, body mass index, blood pressure, haemogram and formula, glycated haemoglobin, total cholesterol, HDL, LDL, triglycerides, albumin, iron, ferritin, vitamin B12, and folate. Adherence to the Mediterranean diet, intervention satisfaction and compliance, and the number of primary care visits will also be measured during pre-intervention (4 months), intervention (4 months), and post-intervention (4 months) periods. Confounding or effect-modifying variables will also be recorded.

Statistical Analysis: Initially, the sociodemographic characteristics of both groups will be described. Percentages will be used for qualitative variables, and means with standard deviations or medians with ranges and interquartile ranges (25-75) for quantitative variables. Baseline scores on selected scales will be compared post-randomisation to ensure no significant differences. Post-intervention, mean scores across scales and variables will be compared for each group independently and for different post-intervention time periods using paired Student's t-tests (for normally distributed data) or Mann-Whitney U tests (for non-normal distributions). Secondary analyses will include multiple regression, incorporating sociodemographic and confounding variables, to assess clinical remission of depression (Yes: Beck scale <12), anxiety (Yes: GAD-7 <10), and social support (Yes: DUKE-UNC-11 >32).

Expected Results:

The intervention group is expected to show improvements in emotional and nutritional status, social support, and quality of life.

Applicability and Relevance:

The proposed solution leverages existing infrastructure-neighbourhood restaurants, historically spaces for gathering and socialisation, which are currently under threat. These venues could become vital players in the socio-health sector, acting as nutrition caretakers for a specific group of individuals. This approach avoids the need for new canteens or facilities, instead relying on skilled professionals who already exist within the community, while also supporting local economic activity.

By enabling individuals experiencing unwanted loneliness to access group dining in pre-trained restaurants, the intervention aims to improve emotional well-being through social interaction, foster better nutrition, and enhance quality of life. These benefits could result in reduced healthcare visits and less need for medication.

DETAILED DESCRIPTION:
ANTECEDENTS:

In Western countries, unwanted loneliness has a prevalence of 24 to 40% among individuals aged 65 and over, and it increases with age (1,2). Correlations have been reported between the feeling of loneliness and various health problems, including mental illnesses such as depression and anxiety, cardiovascular and cerebrovascular diseases, cancer, and low levels of emotional well-being (3,4). The issues caused by loneliness lead to a decline in quality of life, poor disease recovery, increased mortality, and high rates of socio-healthcare resource utilization among older adults (4).

Health-related quality of life (HRQoL) is defined as the perception of the physical, mental, and social effects of illness on well-being (5). HRQoL is considered an important health outcome among the population and an essential public health tool for assessing physical and social functioning, mental health, and well-being, as well as for evaluating population-based intervention programmes (6). Poor HRQoL perceptions have been associated with advanced age, lack of social support, high levels of depression, low self-esteem, lower social class, female gender, chronic medical conditions, high body mass index, and sedentary lifestyles (7).

The percentage of individuals aged 64 and over in Catalonia on 1 January 2023 was 19.34% (1,528,379 individuals) (8), and it is expected to increase further to 26% by 2037, according to data published by the National Institute of Statistics (INE) (9). Promoting quality of life in this population is now a priority for healthcare researchers.

In our society, loneliness, depression, and anxiety are common among older adults. Malnutrition is also a very frequent condition among the elderly and constitutes a significant burden on healthcare and social systems (10).

Loneliness negatively impacts the nutritional status of individuals. Currently, there are programmes within the health and social services system, such as home meal services or social dining facilities, which are prescribed to certain individuals due to mobility, financial, or vulnerability issues. However, there are other groups of "lonely" people who do not receive as much attention regarding their nutrition, and who do not have access to shared spaces that provide balanced meals tailored to their situation, while also facilitating their socialization and encouraging them to leave the house, thus improving their daily activity.

The solution we propose is to leverage existing infrastructure (local or neighbourhood restaurants), which have always been places of gathering and socialization but are currently threatened due to the declining competitiveness of traditional catering. These could become additional agents in the socio-healthcare sector and act as providers of nutrition for a specific group of people. This represents the first innovative point: rather than creating new dining facilities or infrastructure, we aim to preserve valuable existing spaces with skilled professionals, contributing to the economic revitalization of the area.

As mentioned, the most vulnerable individuals are covered by various social or healthcare services, but there is another group at nutritional risk, whose situation will eventually have significant physical and emotional consequences, making them more dependent on the healthcare system, yet currently receive little support. If we consider the aging population's progression, this will be a problem that cannot be solely addressed by the administration. Therefore, if we enable these individuals to access part of their meals in a restaurant (previously trained and with necessary adaptations), we will ensure an improvement in their emotional state through social interaction, leaving the house, and better health. This improvement may result in a reduced need for consultations/visits to healthcare centres for various reasons: they feel cared for and listened to in another environment, their condition (e.g., hypertension, diabetes) is better controlled, requiring less follow-up, etc.

Studying simple, cost-effective strategies that foster synergistic public-private collaboration to create sustainable community networks for healthy eating, autonomy, and socialization, which help improve emotional and nutritional status as well as social relationships, is essential for maintaining the quality of life of individuals experiencing unwanted loneliness.

STUDY HYPOTHESIS Individuals experiencing unwanted loneliness, at risk of anxiety, depression, and malnutrition, will experience improvements in emotional and nutritional status, social support, and quality of life if they attend lunch at a restaurant two or three times a week, in a group, accompanied by a facilitator.

OBJECTIVES (General and Specific)

Main Objective:

• To assess whether attending lunch at a restaurant twice a week, in a group, accompanied by a facilitator, and participating in healthy eating workshops improves emotional and nutritional status, social support, and quality of life for individuals living with unwanted loneliness.

Secondary Objective:

* To understand the perceptions, feelings, and opinions of participants involved in the intervention.
* To study whether the intervention reduces the number of medical visits and prescription medication use.

METHODOLOGY:

* Design: Randomised clinical trial with two groups.
* Study Population: Individuals aged 18 and over enrolled in the basic health area of Sant Joan de Vilatorrada (12,721 enrolled individuals).
* Inclusion Criteria: Autonomous individuals experiencing issues related to living alone or feeling lonely (Z60) (e.g., elderly, migrants, those with functional diversity, etc.), at risk of malnutrition or emotional disorders, with a score of ≥14 and <28 on the Beck Depression Inventory (BDI-II), a score of ≥10 on the Generalized Anxiety Disorder (GAD-7) scale, or a score of ≥32 on the Duke-UNC-11 Social Support Scale; ability to undergo follow-up for 8 months, ability to read and write in Spanish or Catalan, and the ability to attend the restaurant twice a week.
* Exclusion Criteria: Diagnosis of dementia or moderate cognitive impairment, diagnosis of major depression (BDI-II score ≥28), alcohol or drug abuse, physical or mental impairment preventing attendance at the restaurant two or three times a week, failure to sign the informed consent form, participation in other food support programmes by social services, not being responsible for their own nutrition, or lack of economic autonomy to co-finance the service (5 euros per meal).
* Intervention:

The intervention group will dine at a selected and trained restaurant twice a week for 4 months (from March to June 2024). A facilitator will accompany the participants to the restaurant and supervise them. Once a month, a healthy habits and meal supplementation workshop will be held at the senior citizens' centre. Participants will not be required to pay for the meals at the restaurant or for participation in the workshops. The control group will receive standard care at their Primary Care Centre.

In order for the restaurant to provide appropriate services tailored to the users' needs, training will be conducted by professionals from the Alicia Foundation on how to manage the nutrition of elderly individuals and other participants in the study according to their dietary needs.

- Sample Size Calculation: The sample size was determined for independent groups, capable of detecting a 4.5-point difference in the average score of the Beck Depression Inventory (SD of 7 points [1]), a 2.7-point difference in the average score of the GAD-7 scale (SD of 4.5 points [2]), and a 7-point difference on the Duke-UNC-11 Social Support Questionnaire (SD of 10.6 points [3]). One control will be assigned per case, assuming 80% statistical power with a 5% significance level. A 10% dropout rate is expected, and it has been calculated that 49 participants per group, for a total of 98 participants, are required. The GRANMO version 7.12 calculator was used: https://www.imim.es/ofertadeserveis/software-public/granmo (consulted on 15 March 2017).

- Recruitment: Researchers will request the list of patients assigned to the Sant Joan de Vilatorrada Primary Care Centre (CAP) with diagnoses of living alone, related issues (Z60), anxiety (F41), and depression (F32) from the Technical Area of the Central Catalonia Management. The CAP's health and social services will review the list and identify individuals who meet the inclusion criteria. Social services from the local council may also suggest candidates if identified. Once identified, CAP administrative staff, under the guidance of healthcare professionals, will contact them and invite them to participate. If they agree to participate, they will be scheduled for a study explanation, physical examination, blood sample extraction, completion of questionnaires, and informed consent (Annex 1). Their responses will be used to generate the final list of included patients, taking into account the cutoff points of the scales (i.e., BDI-II >14 or GAD >10 or DUKE-UNC-11 >32).

- Group Assignment: Random assignment of patients to the different groups (control and intervention) will be performed using the SPSS statistical programme. Patients with depression, anxiety, and low social support will be equally assigned to the intervention and control groups. Stratified randomization based on age and gender will also be carried out to increase the generalisability of the results.

* Variables and Measurement Methods:

  * Independent Variables:

    o Sociodemographic variables: gender, age, marital status (single, married, separated, widowed), educational level (no formal education, primary education, secondary education, higher education).
  * Dependent Variables:

    * Clinical remission of depression or response to the intervention at the end of the intervention. Clinical remission is defined as a Beck Depression Inventory (BDI-II) score <14, and response to the intervention is defined as a decrease in the initial score [1].
    * Clinical remission of anxiety or response to the intervention at the end of the intervention. Clinical remission is defined as a score <10 on the GAD-7 scale (Generalized Anxiety Disorder), and response to the intervention is defined as a reduction in the baseline score [2].
    * Improvement in social support after the intervention. A response to the intervention is defined by a decrease in the Duke-UNC-11 Social Support Questionnaire score, with a score <32 indicating good social support [3].
    * Improvement in Health-Related Quality of Life (HRQoL) [4,5] after the intervention: an improvement in HRQoL is considered if there is a decrease in the EuroQol (EQ-5D) questionnaire score compared to the baseline.
    * Clinical variables: weight, height, body mass index, blood pressure, complete blood count, haemoglobin A1c, total cholesterol, HDL and LDL cholesterol, triglycerides, albumin, iron, ferritin, vitamin B12, and folate.
    * Adherence to the Mediterranean diet through the validated PREDIMED questionnaire [6].
    * Satisfaction with the intervention: At the end of the intervention, a satisfaction survey will be conducted using a 5-point Likert scale.
    * Adherence to the intervention: Attendance at the restaurant and healthy eating workshops will be recorded. Adherence to the intervention will be calculated as attending 75% or more of the scheduled days.
    * Number of visits made to the primary care centre, emergency department an referrals to the hospital: pre-intervention (4 months), intervention (4 months).
    * Confounding or effect-modifying variables to be considered:
* Pharmacological treatment: The defined daily dose (DDD, WHO) will be calculated for each active component, taking into account the number of days, dispensed dose, and drug administration route. Active ingredients recorded will include those belonging to antidepressant, anxiolytic, antidiabetic, and antihyperlipidemic groups.
* Psychological treatment.

DATA COLLECTION AND SOURCES OF INFORMATION:

Data, both pre- and post-intervention, will be obtained through:

* The previously specified questionnaires.
* Clinical variables: through physical examination and blood extractions. The clinical variables collected for the study are those typically requested during routine check-ups for Primary Care patients.
* Data such as the number of visits during a specified period, prescribed medications, etc., will be extracted through the technical area of the Territorial Management of Central Catalonia.

DATA ANALYSIS:

Initially, the sociodemographic characteristics of both groups will be described. For the description of qualitative variables, percentages will be used, and for quantitative variables, means and standard deviations or means, ranges, and 25th-75th percentiles will be employed.

Prior to the intervention, baseline scores on the selected scales will be compared after randomisation of the patients to ensure no significant differences. Post-intervention, the mean scores of the different scales and variables in both groups will be compared independently, and for the different post-intervention time points, using the Student's t-test for paired samples if the normality assumption holds, or the Mann-Whitney U test if the distribution is not normal. A secondary analysis will be performed using multiple regression, including sociodemographic and confounding variables, for the clinical remission variable of depression (Yes/No) (Yes: Beck scale <12), clinical remission of anxiety (Yes/No) (Yes: GAD-7 <10), and social support (Yes/No) (Yes: DUKE-UNC-11 >32).

Results showing differences with a p-value <0.05 will be considered significant. For statistical analysis, SPSS software version 18 (SPSS Inc., Chicago, IL, USA) will be used.

DIFFICULTIES AND LIMITATIONS OF THE STUDY:

* One potential difficulty will be adherence to the intervention due to the characteristics of the participants: likely elderly individuals, with low social support, and emotional disorders. To mitigate this potential difficulty, the role of the facilitator has been integrated.
* Limitations and barriers in the adoption model: A possible challenge in implementing the project is adapting the restaurant to accommodate specific schedules, diets, and shared tables for users. This adaptation may involve changes to the restaurant's routines and working hours, which could generate resistance or implementation difficulties. To overcome this limitation, close communication and collaboration with participating restaurants will be undertaken to understand their constraints and find appropriate solutions. Joint meetings and working sessions will be held to explore flexible options, such as special hours or adapted menus, that meet the needs and preferences of users while adjusting to the restaurant's existing gastronomic offerings, routines, and staff.
* Limitations and barriers to economic sustainability: Commercialisation, profits, costs, and necessary collaborators are key factors in ensuring the economic sustainability of the solution. This proposal may require stable, adequate funding to cover operational costs, facilitator remuneration, and other related expenses. Efforts will be made to develop a sustainable business model that generates income through various avenues, such as collaboration with participating restaurants, grants, donations, or other available financial resources, as well as the possibility of co-financing the programme by the local government, similar to home meal services.
* Limitations and barriers in coordination: A critical aspect is ensuring efficient coordination and communication among the different stakeholders involved in the project: restaurants, facilitators, healthcare and social professionals, and individuals living alone. Clear protocols, appropriate communication channels, and feedback mechanisms will be established for smooth interaction and effective collaboration.
* Limitations and barriers regarding the necessary collaborators: The implementation of this project requires the collaboration of various actors, such as healthcare staff, local authorities, and third-sector entities. Effective coordination and collaboration with these collaborators are essential for the project's success. Regular meetings will be held, active participation will be encouraged, and communication will be facilitated to ensure smooth collaboration. Mechanisms for recognition and incentives will also be introduced to motivate and reward the participation of key collaborators.

ETHICAL CONSIDERATIONS AND DATA CONFIDENTIALITY Good Clinical Practice Recommendations: This study adheres to the recommendations of Good Clinical Practice, the Declaration of Helsinki of the World Medical Association (revised at the 64th General Assembly, Fortaleza, Brazil, October 2013), and applicable legal regulations.

Participant Information and Types of Consent Requested: Participants will be informed about the study verbally by one of the researchers and through the participant information sheet. If they agree to participate, they will be asked to voluntarily sign the Informed Consent form (Appendix 1).

Data Processing and Confidentiality: It is guaranteed that the strictest professional conduct and confidentiality standards will be maintained at all times, in compliance with Regulation (EU) 2016/679 of the European Parliament and the Council of 27 April 2016 on the protection of natural persons (GDPR) and Organic Law 3/2018, of 5 December, on the Protection of Personal Data and the Guarantee of Digital Rights (LOPD-GDD). The participant's right to confidentiality is paramount. The participant's identity in study documents will be coded, and only authorised personnel will have access to identifiable personal details if data verification processes require inspection of those details. Identifiable personal details will therefore remain confidential at all times and will only be accessible to the Principal Investigator (PI) and authorised personnel.

The data collected will be kept for five years to ensure the integrity of the study, the replicability of the results, and the verification of the conclusions, as well as to be available for any future consultations, verifications, or publications related to the results.

Data will not be transferred to third parties outside the research team, and no international transfers are anticipated. Adequate security measures will be ensured to prevent breaches of confidentiality and privacy. The ICS takes responsibility and guarantees the protection of data storage, preservation, and processing, ensuring confidentiality. Data will be collected through paper questionnaires and, along with the informed consents, stored at the ICS's USR of Central Catalonia, under the custody of the PI. ICS will be responsible for the data processing, and the PI will use the data responsibly. Paper-based data will be linked to a patient code, and a coded database in Excel format will be created and stored on ICS servers with a password, where only the Principal Investigator will have access.

Upon completion of the study, the research team reserves the right to exploit the database for scientific purposes (research articles, working scientific documents, and book chapters).

The researchers declare no conflict of interest. This project has been evaluated by the Ethics Committee of IDIAP Jordi Gol, under code 23/285-P

APPLICABILITY AND PRACTICAL UTILITY OF THE STUDY RESULTS Loneliness has a negative impact on the nutritional status of individuals. Currently, there are programs provided by social and healthcare services within the health system or municipalities, such as home meal delivery services or social dining facilities, which are prescribed to certain individuals due to mobility issues, financial difficulties, or significant vulnerability. However, there are other groups of "lonely" individuals whose nutritional needs are not as closely monitored, and who do not have access to shared spaces that provide balanced meals tailored to their situation, while also facilitating socialisation and encouraging them to leave their homes, thus improving their daily activity.

The solution we propose is to make use of existing infrastructures (local or neighbourhood restaurants), which have historically served as spaces for gathering and socialisation, and which are currently under threat due to the increasing uncompetitiveness of traditional restaurants. These establishments could become an additional agent in the socio-health sector, acting as caregivers for the nutrition of a specific group of individuals. This is an innovative first step: instead of creating new dining halls or new infrastructures, we aim to utilise spaces that already exist, with skilled professionals we wish to preserve, while also promoting the economic revitalisation of a territory.

As previously mentioned, the most vulnerable individuals are covered by various social or healthcare services, but there is another group at risk of poor nutrition, a condition that will eventually have significant physical and emotional consequences, making them more dependent on the healthcare system, yet currently receiving little support. Considering the progression of population ageing, this will be a problem that will be difficult to address solely by the administration.

Therefore, if we enable these individuals to access some of their meals in a restaurant (previously trained and appropriately adapted), we can ensure an improvement in their emotional state due to social interaction, leaving their homes, and improving their health status. This improvement may result in a reduced need for healthcare visits for various reasons: they feel cared for and listened to elsewhere, their condition (hypertension, diabetes, etc.) is better controlled, requiring less follow-up, etc.

The proposed solution seeks to establish mechanisms and create an ecosystem through which healthcare and social services can prescribe dining at a restaurant (pre-selected and trained to be part of the network offering this service) at a determined frequency, allowing for socialisation without stigmatisation and without the need to create new infrastructures or hire additional staff.

AVAILABLE RESOURCES FOR PROJECT IMPLEMENTATION Grant from the First Call of the Social and Healthcare Innovation Hub (HiSS), the challenge of Unwanted Loneliness.

JUSTIFICATION FOR THE REQUESTESD LONELINESS The requested funding is necessary to launch a pilot programme in the town of Sant Joan de Vilatorrada, a municipality in the Bages region, which already has an established network in community health. Social and healthcare services will prescribe that a group of individuals living in unwanted loneliness attend a pre-selected restaurant trained in healthy eating. Participants, accompanied by a facilitator, will not only receive sufficient and balanced meals at the restaurants but will also have a space to promote socialisation and education through healthy eating workshops.

This grant is requested to cover:

1. The hours of professionals dedicated to the project (coordination, recruitment, data collection, training for restaurant staff, educational sessions for users, etc.).
2. Hiring staff to carry out specific tasks during the proof of concept (facilitator).
3. Funding for impact evaluation and any potential resulting publications.
4. Covering costs associated with the participating restaurants.
5. The preparation of educational materials.
6. Transport expenses.

The professionals involved in the project to varying degrees will include:

* Specialists in nutrition, food, cooking, and food culture from the Alícia Foundation.
* Primary Care research experts and researchers from IDIAP Jordi Gol.
* Professionals from the healthcare and social services in Sant Joan de Vilatorrada.

ELIGIBILITY:
Inclusion Criteria:

* Autonomous individuals experiencing issues related to living alone or feeling lonely (Z60) (e.g., elderly, migrants, those with functional diversity, etc.), at risk of malnutrition or emotional disorders, with a score of ≥14 and <28 on the Beck Depression Inventory (BDI-II), a score of ≥10 on the Generalized Anxiety Disorder (GAD-7) scale, or a score of ≥32 on the Duke-UNC-11 Social Support Scale; ability to undergo follow-up for 8 months, ability to read and write in Spanish or Catalan, and the ability to attend the restaurant twice a week.

Exclusion Criteria:

* Diagnosis of dementia or moderate cognitive impairment, diagnosis of major depression (BDI-II score ≥28), alcohol or drug abuse, physical or mental impairment preventing attendance at the restaurant two or three times a week, failure to sign the informed consent form, participation in other food support programmes by social services or not being responsible for their own nutrition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Depression | 4 months
  Clinical remission of depression or response to the intervention at the end of the intervention. Clinical remission is defined as a Beck Depression Inventory (BDI-II) score <14, and response to the intervention is defined as a decrease in the initial score
Anxiety | 4 months
  Clinical remission of anxiety or response to the intervention at the end of the intervention. Clinical remission is defined as a score <10 on the GAD-7 scale (Generalized Anxiety Disorder), and response to the intervention is defined as a reduction in the baseline score
Social support | 4 months
  Improvement in social support after the intervention. A response to the intervention is defined by a decrease in the Duke-UNC-11 Social Support Questionnaire score, with a score <32 indicating good social support
Health-Related Quality of Life | 4 months
  Improvement in Health-Related Quality of Life (HRQoL) after the intervention: an improvement in HRQoL is considered if there is a decrease in the EuroQol (EQ-5D) questionnaire score compared to the baseline.

SECONDARY OUTCOMES:
Clinical variables | 4 months
  weight, height, body mass index, blood pressure, complete blood count, haemoglobin A1c, total cholesterol, HDL and LDL cholesterol, triglycerides, albumin, iron, ferritin, vitamin B12, and folate
Adherence to the Mediterranean diet | 4 months
  Adherence to the Mediterranean diet through the validated PREDIMED questionnaire
Visits made to the primary care centre | 8 months
  Number of visits made to the primary care centre: pre-intervention (4 months), intervention (4 months)
Visits made to the emergency department | 8 months
  Number of visits made to the emergency department: pre-intervention (4 months), intervention (4 months), post-intervention (4 months).
Referrals to the hospital | 8 months
  Number of referrals to the hospital: pre-intervention (4 months), intervention (4 months)
Satisfaction with the intervention | 4 months
  Satisfaction with the intervention: At the end of the intervention, a satisfaction survey will be conducted using a 5-point Likert scale
Adherence to the intervention | 4 months
  Adherence to the intervention: Attendance at the restaurant and healthy eating workshops will be recorded. Adherence to the intervention will be calculated as attending 75% or more of the scheduled days.

CONTACTS AND LOCATIONS:
Locations (1):
- Unitat de Suport a la Recerca de la Catalunya Central, Fundació Institut Universitari per a la Recerca a l'Atenció Primària de Salut Jordi Gol i Gurina, Manresa, Spain, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rockwood K. What would make a definition of frailty successful? Age Ageing. 2005 Sep;34(5):432-4. doi: 10.1093/ageing/afi146. PMID 16107450
- [Background] Urzua M A. [Health related quality of life: Conceptual elements]. Rev Med Chil. 2010 Mar;138(3):358-65. Epub 2010 May 19. Spanish. PMID 20556342
- [Background] 8. Institut d'Estadística de Catalunya. Població a 1 de gener 2023. Available online: https://www.idescat.cat/indicadors/?id=aec&n=15231 (accessed on 24 october 2023).Proyecciones de Población 2022-2072. Available online: https://www.ine.es/prensa/pp_2022_2072.pdf (accessed on 24 october 2023).
- [Background] Gene-Badia J, Comice P, Belchin A, Erdozain MA, Caliz L, Torres S, Rodriguez R. [Profiles of loneliness and social isolation in urban population]. Aten Primaria. 2020 Apr;52(4):224-232. doi: 10.1016/j.aprim.2018.09.012. Epub 2019 Feb 12. Spanish. PMID 30770152
- [Background] Lubetkin EI, Jia H, Franks P, Gold MR. Relationship among sociodemographic factors, clinical conditions, and health-related quality of life: examining the EQ-5D in the U.S. general population. Qual Life Res. 2005 Dec;14(10):2187-96. doi: 10.1007/s11136-005-8028-5. PMID 16328899
- [Background] Dent E, Wright ORL, Woo J, Hoogendijk EO. Malnutrition in older adults. Lancet. 2023 Mar 18;401(10380):951-966. doi: 10.1016/S0140-6736(22)02612-5. Epub 2023 Jan 27. PMID 36716756
- [Background] Cacioppo JT, Cacioppo S. Older adults reporting social isolation or loneliness show poorer cognitive function 4 years later. Evid Based Nurs. 2014 Apr;17(2):59-60. doi: 10.1136/eb-2013-101379. Epub 2013 Jun 8. No abstract available. PMID 23749730
- [Background] Nyqvist F, Nygard M, Scharf T. Loneliness amongst older people in Europe: a comparative study of welfare regimes. Eur J Ageing. 2018 Sep 6;16(2):133-143. doi: 10.1007/s10433-018-0487-y. eCollection 2019 Jun. PMID 31139028